CLINICAL TRIAL: NCT06141018
Title: Safety and Effectiveness of Intra-articular Injection of a Cross-linked Sodium Hyaluronate in Knee Osteoarthritis: A Randomized, Prospective, Double-blind, Placebo-controlled, Cross-over, Post-marketing Clinical Follow-up Study
Brief Title: Effectiveness and Safety of Intra-articular SEMICAL GEL-B CROSS Therapy in Knee Osteoarthritis (SEM-ART1)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semikal Technology (Industry)
Collaborators: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SEM-ART1
Record Dates: First submitted 2023-10-25; First posted 2023-11-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; hyaluronic acid; intraarticular injection; viscosupplementation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cross-linked intra-articular hyaluronic acid (Active Comparator): Cross-linked intra-articular hyaluronic acid (90 mg 3 ml cross-linked hyaluronic acid)
  Interventions: Device: Cross-linked intra-articular hyaluronic acid
- Placebo (Placebo Comparator): Intra-articular isotonic saline solution (3 ml 0.9% isotonic saline) at the same dose as the treatment arm
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Cross-linked intra-articular hyaluronic acid — Patients in the treatment arm will receive 3 ml, 90 mg hyaluronic acid injection intra-articularly, while the ones in the placebo arm will receive 3 ml saline injection intra-articularly. The groups will be crossed-over at 3rd month.
  Arms: Cross-linked intra-articular hyaluronic acid
Other: Placebo — Patients in the treatment arm will receive 3 ml, 90 mg hyaluronic acid injection intra-articularly, while the ones in the placebo arm will receive 3 ml saline injection intra-articularly. The groups will be crossed-over at 3rd month.
  Other Names: 3 ml isotonic saline solution
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of intra-articular injection of a cross-linked sodium hyaluronate; SEMICAL GEL-B CROSS, in knee osteoarthritis.

Primary objectives: The aim of this study is to obtain short- and long-term clinical data on the performance and safety of intra-articular injection of SEMICAL GEL B-CROSS, produced and marketed by Semical Biosurgery incorporated company, in knee osteoarthritis patients.

It is also aimed to monitoring known adverse events and complications, detecting previously unknown adverse events and complications, to identify and analyze emerging risks based on real-life data. Participants will receive intra-articular injection of either a cross-linked sodium hyaluronate (SEMICAL GEL-B CROSS); or placebo (isotonic saline solution) at baseline, and will be followed-up for one year to compare the effectiveness and safety of the given therapy.

DETAILED DESCRIPTION:
The study is a randomized controlled, double-blind, two-armed, single-center and cross-over study. After a maximum screening period of 28 days, patients with Kellgren & Lawrence Stage II and III knee osteoarthritis will be randomly assigned to one of the two treatment arms on the day of injection, which is considered Day 0. These treatment arms are:

Group 1: Treatment Arm - Cross-linked intra-articular hyaluronic acid (90 mg 3 ml cross-linked hyaluronic acid)

Group 2: Control Arm - Intra-articular isotonic saline solution (3 ml 0.9% isotonic saline) A safety visit will be made 7-10 days after administration of the treatment injection and the injection site will be visually evaluated for local reactions. In addition, an inquiry for injection-related adverse events will also be conducted.

Treatment responses of patients in both groups will be evaluated by a separate researcher blinded to study treatment with predefined objective response criteria.

At the 3rd month visit, the patients in both groups will be crossed-over and those who received a placebo at baseline will receive a hyaluronic acid injection at the 3rd month, while those who receive a hyaluronic acid injection at baseline will receive a placebo at the 3rd month. Efficacy evaluations will continue to be made at every three months for one year.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over, both male and female
* Diagnosed with clinical knee osteoarthritis according to the American College of
* Rheumatology (ACR) criteria, with Kellgren & Lawrence stage II and III osteoarthritic findings on antero-posterior knee radiographs
* Able to provide written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain scores | Baseline, 3 months, 6 months, 9 months, and 12 months.
  The alteration in pain arising from knee osteoarthritis will be assessed in correlation with changes in WOMAC pain scores at baseline, 3 months, 6 months, 9 months, and 12 months.

SECONDARY OUTCOMES:
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) function score | Baseline, 3 months, 6 months, 9 months, and 12 months.
  The alteration in pain arising from knee osteoarthritis will be assessed in correlation with changes in WOMAC pain scores at baseline, 3 months, 6 months, 9 months, and 12 months.
Changes in knee functions | Baseline, 3 months, 6 months, 9 months, and 12 months.
  The alteration in function arising from knee osteoarthritis will be assessed in correlation with changes in WOMAC pain scores at baseline, 3 months, 6 months, 9 months, and 12 months.
Changes in knee flexor muscle strength | Baseline, 3 months, 6 months, 9 months, and 12 months.
  Knee flexor muscle strength assessed by myometer
Changes in knee extensor muscle strength | Baseline, 3 months, 6 months, 9 months, and 12 months.
  Knee extensor muscle strength assessed by myometer
Changes in knee functions during 5 times sit to stand test | Baseline, 3 months, 6 months, 9 months, and 12 months.
  5 times sit to stand test
Changes in knee functions by 6MWT (6 Minute Walking Test) | Baseline, 3 months, 6 months, 9 months, and 12 months.
  6 minute walking test
Change in the need for analgesic drug from pre-treatment to post-treatment | Baseline, 3 months, 6 months, 9 months, and 12 months.
  Will be assessed by patient diary
Change in quality of life | Baseline, 3 months, 6 months, 9 months, and 12 months.
  Will be assessed by 36-item Short Form Survey
Change in knee pain during movement and rest | Baseline, 3 months, 6 months, 9 months, and 12 months.
  Will be assessed by Visual Analogue Scale 1-10 (1: no pain, 10: very much pain)
Local reactions in the injection site | 7-10 days post-injection
  A safety visit will be performed 7-10 days after administration of the treatment injection and the injection site will be visually assessed for local reactions.
Adverse events throughout the entire study period | Through study completion, an average of 1 year.
  Adverse events will be questioned throughout the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Kara, Study Director — Semikal Technology
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol will be published as an article.